CLINICAL TRIAL: NCT00455572
Title: Cancer Immunotherapeutic GSK1572932A as Adjuvant Therapy for Patients With MAGE-A3-positive Non-Small Cell Lung Cancer
Brief Title: Cancer Immunotherapy GSK1572932A as Adjuvant Therapy for Patients With Tumor-antigen-positive Non-Small Cell Lung Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study early termination was due to slow recruitment and difficulties at achieving the required enrolment for the study.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 107240
Record Dates: First submitted 2007-04-02; First posted 2007-04-03 (Estimated); Last update posted 2017-05-15 (Actual); Status verified 2017-05

CONDITIONS: Lung Cancer, Non-Small Cell
Keywords: Immunotherapeutic; Adjuvant cancer therapy; Non-small-cell lung cancer; ASCI
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Cisplatin; Vinorelbine; Radiotherapy

ARMS (4):
- Cohort 1 (Experimental): Patients with resected stage IB, II or IIIA tumors who are due for standard chemotherapy with cisplatin and vinorelbine. These patients will receive chemo-and immunotherapy in parallel.
  Interventions: Biological: Immunotherapeutic GSK1572932A; Drug: Cisplatin (CDDP); Drug: Vinorelbine
- Cohort 2 (Experimental): Patients with resected stage IB, II or IIIA tumors who are due for standard chemotherapy with cisplatin and vinorelbine. These patients will first receive chemotherapy and then immunotherapy
  Interventions: Biological: Immunotherapeutic GSK1572932A; Drug: Cisplatin (CDDP); Drug: Vinorelbine
- Cohort 3 (Experimental): Patients with resected stage IB, II or IIIA tumors who are not due for chemotherapy. These patients will receive immunotherapy only.
  Interventions: Biological: Immunotherapeutic GSK1572932A
- Cohort 4 (Experimental): Patients with unresectable stage III tumors, following standard chemotherapy and/or radiotherapy. These patients will receive immunotherapy only.
  Interventions: Biological: Immunotherapeutic GSK1572932A; Drug: Cisplatin (CDDP); Drug: Vinorelbine; Procedure: Radiotherapy

INTERVENTIONS:
Biological: Immunotherapeutic GSK1572932A — Intramuscular injection, 8 doses
Drug: Cisplatin (CDDP) — Four cycles with doses based on patient's body surface area, intravenous administration
  Arms: Cohort 1; Cohort 2; Cohort 4
Drug: Vinorelbine — Four cycles with doses based on patient's body surface area , intravenous administration
  Arms: Cohort 1; Cohort 2; Cohort 4
Procedure: Radiotherapy — Regimen will be based upon the site's own standard procedures
  Arms: Cohort 4

SUMMARY:
The purpose of this clinical trial is to find out how successfully non-small-cell lung cancer patients are able to give an immune response to injections of the immunotherapeutic product GSK1572932A, and to find out more about the safety of this treatment. A course of eight injections will be administered over 21 weeks; including screening for suitability and all tests, the duration of the study for a patient will be 30-35 weeks. During this period various tests will be performed, including physical examinations and blood tests. The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007.

DETAILED DESCRIPTION:
This is an open, four-arm, parallel-group study, to be conducted at approximately 20 centers in Europe and Canada. All patients will receive the same immunotherapeutic treatment with GSK1572932A, but they will be recruited into four cohorts according to the details of their disease. Cohort 1: Patients with resected stage IB, II or IIIA tumors who are due for standard chemotherapy with cisplatin and vinorelbine. These patients will receive chemo-and immunotherapy in parallel. Cohort 2: Patients with resected stage IB, II or IIIA tumors who are due for standard chemotherapy with cisplatin and vinorelbine. These patients will first receive chemotherapy and then immunotherapy.

Cohort 3: Patients with resected stage IB, II or IIIA tumors who are not due for chemotherapy. These patients will receive immunotherapy only. Cohort 4: Patients with unresectable stage III tumors, following standard chemotherapy and/or radiotherapy. These patients will receive immunotherapy only. Immunotherapeutic treatment will comprise eight doses of GSK1572932A. Doses will be administered at three-week intervals; in Cohort 1 this may be adapted to fit in with the patient's chemotherapy. During the study, adjuvant radiotherapy is allowed in Cohorts 1, 2 and 3 for patients in stage III only and is prohibited in Cohort 4. Chemotherapy during the study is allowed in Cohort 1 only as described above, and is prohibited in Cohorts 2-4. The total maximum duration of the study for a patient will be 30-35 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained,
* Aged 18 or more,
* Pathologically proven stage IB, II or III NSCLC,
* Tumor expresses MAGE-A3,
* Free of distant metastasis,
* For Cohort 1, all of the following:

  1. Completely resected stage IB, II or IIIA NSCLC,
  2. Anatomical tumor resection, involving at least a lobectomy, and nodal sampling as per center standard
  3. ECOG performance status = 0 or 1
  4. Due to receive adjuvant chemotherapy as permitted in the protocol
  5. Not received, not receiving, and not due to receive adjuvant radiotherapy (except stage III patients)
  6. First administration of chemotherapy can be scheduled within 4-12 weeks after surgery
* For Cohort 2, all of the following:

  1. Resected stage IB, II or IIIA NSCLC,
  2. Anatomical tumor resection, involving at least a lobectomy, and nodal sampling as per center standard
  3. ECOG PS = 0 or 1
  4. Due to receive, or receiving, adjuvant chemotherapy as permitted in the protocol
  5. Not received, not receiving, and not due to receive, adjuvant radiotherapy (except stage III patients)
  6. First administration of ASCI treatment can be scheduled within 2-4 weeks after the last administration of chemotherapy
  7. Received at least 2 cycles of standard chemotherapy before ASCI treatment is initiated, whereafter no further chemotherapy is planned
* For Cohort 3, all of the following:

  1. Resected stage IB, II or IIIA NSCLC
  2. Anatomical tumor resection, involving at least a lobectomy, and nodal sampling as per center standard
  3. ECOG PS = 0 or 1 or 2
  4. Not received, not receiving, and not due to receive, adjuvant chemotherapy
  5. Not received, not receiving, and not due to receive, adjuvant radiotherapy (this does not apply to patients in stage III)
  6. First administration of ASCI treatment can be scheduled within 4-8 weeks after surgery
* For Cohort 4, all of the following:

  1. Unresectable stage III NSCLC
  2. ECOG PS = 0 or 1 or 2
  3. Due to receive, or receiving, chemo- and radiotherapy according to institution standard
  4. Received at least 2 cycles of standard chemotherapy before the initiation of ASCI treatment, whereafter no further chemo-/radiotherapy is planned
  5. Stable disease or objective response (confirmed by CT scan) after standard chemo-/radiotherapy
  6. Administration of ASCI treatment can be scheduled within 2-6 weeks after the last administration of chemo-/radiotherapy
* Laboratory criteria: adequate bone-marrow reserve, adequate renal function, adequate hepatic function.
* For females: EITHER not of child-bearing potential, OR sexually abstinent, OR negative urine pregnancy test + use of adequate contraceptive precautions from 30 days before first study treatment till 2 months after completion of study treatment course
* In the view of the investigator, the patient can and will comply with the requirements of the protocol

Exclusion criteria:

* Previous or concomitant other malignancies, except if effectively treated and considered by the investigator highly likely to have been cured
* Pregnant or lactating
* History of anaphylaxis or severe allergic reaction
* Concurrent severe medical problems, unrelated to the malignancy, limiting full compliance with the study or exposing the patient to unacceptable risk
* Psychiatric or addictive disorders compromising the ability to give informed consent, or to comply with the trial procedures
* HIV-positive
* Require treatment with systemic corticosteroids, or other immunosuppressive agents
* Need home oxygenation
* Received or plan to receive investigational or non-registered product other than the study medication from 30 days before first dose of study medication and during whole study period
* History of chronic alcohol consumption and/or drug abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2007-05-11 (Actual); Primary Completion 2013-08-04 (Actual); Study Completion 2013-08-08 (Actual)

PRIMARY OUTCOMES:
The anti-MAGE-A3 seroconversion | After the fourth dose of ASCI and at the end of treatment
The anti-protein D seroconversion | After the fourth dose of ASCI and at the end of treatment
The anti-CpG seroconversion | After the fourth dose of ASCI and at the end of treatment
The MAGE-A3 cellular (T cell) response | After the fourth dose of ASCI and at the end of treatment
Occurrence of adverse events, including abnormal hematological and biochemical laboratory values | During the study
Occurrence of serious adverse events | During the study

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (25):
- Belgium (3):
  - GSK Investigational Site, Genk
  - GSK Investigational Site, Leuven
  - GSK Investigational Site, Liège
- Canada (3):
  - GSK Investigational Site, Edmonton, Alberta
  - GSK Investigational Site, Greenfield Park, Quebec
  - GSK Investigational Site, Montreal, Quebec
- France (4):
  - GSK Investigational Site, Montpellier
  - GSK Investigational Site, Pierre-Bénite
  - GSK Investigational Site, Saint-Herblain
  - GSK Investigational Site, Strasbourg
- Germany (6):
  - GSK Investigational Site, Hemer, North Rhine-Westphalia
  - GSK Investigational Site, Mainz, Rhineland-Palatinate
  - GSK Investigational Site, Halle, Saxony-Anhalt
  - GSK Investigational Site, Großhansdorf, Schleswig-Holstein
  - GSK Investigational Site, Bad Berka, Thuringia
  - GSK Investigational Site, Hamburg
- Italy (4):
  - GSK Investigational Site, Udine, Friuli Venezia Giulia
  - GSK Investigational Site, Rome, Lazio
  - GSK Investigational Site, Genoa, Liguria
  - GSK Investigational Site, Milan, Lombardy
- United Kingdom (5):
  - GSK Investigational Site, Wythenshawe, Greater Manchester
  - GSK Investigational Site, Bebington, Wirral
  - GSK Investigational Site, London
  - GSK Investigational Site, Nottingham
  - GSK Investigational Site, Southampton

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Pujol JL, Vansteenkiste JF, De Pas TM, Atanackovic D, Reck M, Thomeer M, Douillard JY, Fasola G, Potter V, Taylor P, Bosquee L, Scheubel R, Jarnjak S, Debois M, de Sousa Alves P, Louahed J, Brichard VG, Lehmann FF. Safety and Immunogenicity of MAGE-A3 Cancer Immunotherapeutic with or without Adjuvant Chemotherapy in Patients with Resected Stage IB to III MAGE-A3-Positive Non-Small-Cell Lung Cancer. J Thorac Oncol. 2015 Oct;10(10):1458-67. doi: 10.1097/JTO.0000000000000653. PMID 26309191
- See also: Results for study 107240 can be found on the GSK Clinical Study Register — https://www.gsk-clinicalstudyregister.com/study/107240?search=study&b%22b''%22#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: 107240 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 107240 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 107240 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 107240 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 107240 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 107240 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 107240 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register